CLINICAL TRIAL: NCT01954498
Title: Effect of Walnuts on Sperm Parameters and Male Fertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Wendie A Robbins, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20130929
Record Dates: First submitted 2013-09-20; First posted 2013-10-01 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Oligozoospermia; Asthenozoospermia; Teratozoospermia; Fertility
Keywords: Randomized controlled trial; Spermatozoa; Sperm; Male Infertility; Walnuts; Nutrition; Male Reproduction
MeSH Terms: conditions — Oligospermia; Asthenozoospermia; Teratozoospermia; Infertility, Male

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walnuts (Experimental): 2 ounces whole-shelled walnuts per day for 12 weeks
  Interventions: Dietary Supplement: Walnuts
- OTC (over-the-counter) multivitamin (Active Comparator): OTC multivitamin tablet 2 per day for 12 weeks
  Interventions: Dietary Supplement: OTC multivitamin

INTERVENTIONS:
Dietary Supplement: Walnuts
  Arms: Walnuts
Dietary Supplement: OTC multivitamin
  Arms: OTC (over-the-counter) multivitamin

SUMMARY:
The investigators are testing the hypothesis that two ounces of whole-shelled walnuts/day added to the diet of men seeking care for infertility will beneficially affect sperm parameters and fertility. The investigators will compare the walnut intervention to the commonly suggested recommendation of adding an OTC multivitamin supplement to the diet.

DETAILED DESCRIPTION:
Purpose: The investigators are testing the hypothesis that two ounces of whole-shelled walnuts/day added to the diet of men with oligo- astheno- or teratospermia will beneficially affect sperm parameters. The investigators found in a previous study (Robbins et al. 2012, Biology of Reproduction 87(4):101, 1-8.) that walnuts added to a Western diet improved sperm parameters in healthy, young men of unknown fertility and the most improvement occurred in participants with poor sperm parameters at baseline. The investigators now test the walnut dietary intervention in a fertility clinic population known to have poor sperm parameters. The investigators will compare the walnut intervention to the usual care suggestion of adding an OTC multivitamin supplement to the diet. Neither walnuts nor the OTC multivitamin have been tested for efficacy in this fertility clinic population previously.

Methods: A randomized, parallel two-group, dietary intervention trial with single-blind masking of outcome assessors will be conducted with up to 140 men who present for fertility work-up with semen parameters below the 25th centile for count, and 10th centile for motility and/or morphology according to the WHO 5th Edition, Laboratory Manual for the Processing and Examining of Human Semen, 2010. Repeated measures at baseline and 12 weeks include: semen analyses (primary outcome), blood fatty acid/ nutrient profiles (secondary outcomes); IPAQ physical activity questionnaire and IIEF index of erectile function (potential modifiers or confounders). Dietary intake will be assessed throughout using 24-hour ASA dietary recall x 5 and fertility assessed by questionnaire at one year post enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older
* Sperm concentration < or = to 41 million per ml
* Sperm motility < or = to 40%
* Normal sperm morphology forms < or = to 5.5%
* Patients of Howard H. Kim, MD seen at the Male Reproductive Medicine and Microsurgery Clinic, Cedars-Sinai Medical Center, Los Angeles, California
* Have eaten walnuts throughout life without adverse reaction

Exclusion Criteria:

* Allergy to walnuts or tree nuts
* Food allergy
* Known genetic cause of infertility
* Known anatomical cause of infertility
* History of seizure disorder

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Sperm count | 12 weeks
  Change from baseline to three months in sperm count
Sperm motility | 12 weeks
  Change from baseline to 12 weeks in sperm motility
Sperm morphology | 12 weeks
  Change from baseline to 12 weeks in sperm morphology

SECONDARY OUTCOMES:
Fertility | 12 months
  Fertilization of ova through natural conception or assisted reproductive technology
Blood fatty acid and nutrient profile | 12 weeks
  Change from baseline to 12 weeks in blood fatty acid profile and nutrients
Sperm aneuploidy | 12 weeks
  Change from baseline to 12 weeks in sperm aneuploidy
Sperm DNA strand breakage | 12 weeks
  Change from baseline to 12 weeks in sperm DNA integrity

OTHER OUTCOMES:
Physical Activity | 12 weeks
  IPAQ (International Physical Activity Questionnaire) assessment of change from baseline to 12 weeks
Sexual function | 12 weeks
  IIEF (International Index of Erectile Function) assessment of change from baseline to 12 weeks
Dietary intake | 12 weeks
  ASA-24 (Automated Self-administered) 24-hour dietary recalls x 5 over 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Howard H Kim, MD, Principal Investigator — Cedars-Sinai Medical Center, Los Angeles, CA; Wendie A Robbins, RN, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Male Reproductive Medicine and Microsurgery Clinic, Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California

REFERENCES:
- [Background] Robbins WA, Xun L, FitzGerald LZ, Esguerra S, Henning SM, Carpenter CL. Walnuts improve semen quality in men consuming a Western-style diet: randomized control dietary intervention trial. Biol Reprod. 2012 Oct 25;87(4):101. doi: 10.1095/biolreprod.112.101634. Print 2012 Oct. PMID 22895856